CLINICAL TRIAL: NCT03760354
Title: Corticosteroid Treatment in the Acute Phase of Caustic Ingestion Management for the Prevention of Refractory Stenosis of the Esophagus and Pharynx- The CORTICAU Study
Brief Title: Corticosteroid Treatment in the Acute Phase of Caustic Ingestion Management
Acronym: CORTICAU
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P160803-J
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Caustic Esophageal Injury; Esophageal Stenosis; Pharyngeal Stenosis
Keywords: Caustic; Esophageal Stenosis; Pharyngeal Stenosis; Corticosteroid treatment
MeSH Terms: conditions — Esophageal Stenosis | interventions — Methylprednisolone

STUDY DESIGN:
Intervention Model Description: Prospective Phase II, Bayesian, single-blinded, monocentric, randomized, prospective clinical trial
Who Masked: Participant
Masking Description: single-blinded trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone (Experimental): Dose: 500mg/day for the first two days then 2mg/kg per day for three days. Dilution in 0.9% NaCl, 100 ml as a single slow intravenous administration over 60 minutes Total processing time of 5 days
  Interventions: Drug: Methylprednisolone
- Placebo (no corticosteroid treatment) (Placebo Comparator): NaCl 0.9%, 100ml per day as a single slow intravenous administration over 60 minutes for a total treatment duration of 5 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Methylprednisolone — Dose: 500mg/day for the first two days then 2mg/kg per day for three days. Dilution in 0.9% NaCl, 100 ml as a single slow intravenous administration over 60 minutes Total processing time of 5 days
  Other Names: Corticosteroid treatment
  Arms: Methylprednisolone
Other: Placebo — NaCl 0.9%, 100ml per day as a single slow intravenous administration over 60 minutes for a total treatment duration of 5 days
  Other Names: Control Arm
  Arms: Placebo (no corticosteroid treatment)

SUMMARY:
The management of patients who have ingested a caustic product has changed since 2007. Whereas previously the lesion assessment and surgical indication were based on endoscopic data, the therapeutic algorithm is currently based solely on the results of a CT scan with contrast injection, performed 6 hours after ingestion. This examination makes it possible to reliably assess the viability of the esophageal and gastric walls and thus to indicate digestive resection. The therapeutic consequences of this new treatment are important because, by expanding the indications for conservative treatment after severe ingestion, it brings a significant gain in terms of survival, morbidity and functional outcome. In the absence of emergency digestive resection, however, the functional prognosis is often overshadowed by the formation of esophageal stenosis in the months following ingestion. Patients then require endoscopic dilation treatment. In the event of failure or impossibility of dilation, which defines refractory stenosis, esophageal reconstruction is necessary. In case of sequential pharyngeal stenosis following ingestion, esophageal and pharyngeal reconstruction is indicated as a first-line treatment, since these stenosis do not respond to endoscopic dilations. The expansion of the indications for conservative treatment after severe ingestion using CT scans has led to an increase in the incidence of after-effect stenosis.

We aim to develop a therapeutic approach that will prevent the development of refractory and pharyngeal esophageal stenosis. Indeed, there is currently no strategy that has proven effective in this regard in adults. The value of corticosteroid therapy for the prevention of caustic stenosis has only been evaluated in children and remains controversial.

The main objective is to evaluate the effect of early systemic corticosteroid therapy on the risk of refractory esophageal or pharyngeal stenosis within one year of ingestion of a caustic substance in a population of patients at high risk of stenosis, defined according to tomodensitometric criteria (grade IIb: severe lesions, absence of transparietal necrosis), and for whom there is no indication of urgent digestive resection.

ELIGIBILITY:
Inclusion Criteria

* Age greater than or equal to 18 years
* Recent caustic product ingestion (time between taking the product and initiating the evaluated treatment or placebo between 6 and 24 hours after ingestion)
* Predictive CT criteria for high-risk esophageal stenosis (grade IIb) in its most pathological part
* Written, signed consent (trusted person if necessary, in case of impossibility of collection)
* Beneficiary of a social security system

Exclusion Criteria:

* Indication of resection or surgical exploration in emergency
* History of caustic ingestion
* Corticosteroids taken at a dose greater than 20 mg prednisone within 7 days before randomization
* Contraindication to corticosteroid therapy:
* Any infectious condition that required antibiotic treatment within 7 days of randomization
* Any vaccine living within 7 days of randomization
* Hypersensitivity to one of the components
* Pregnancy in progress
* Breastfeeding in progress
* Co-intoxication involving vital prognosis and requiring, according to the patient's doctor, intensive care management
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-15 (Estimated); Primary Completion 2020-02-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Indication for esophageal or pharyngeal surgical reconstruction | within 12 months post ingestion
  The primary outcome is the indication for esophageal or pharyngeal surgical reconstruction due to:
  1. The occurrence of one or more esophageal stenosis refractory to endoscopic dilation within 12 months of ingestion, as defined by:
     * The need for more than 5 sessions of esophageal endoscopic dilation
     * Non-expandable stenosis or esophageal obstruction;
     * An esophageal perforation that occurs during dilation, which contraindicates the continuation of dilation.
  2. The occurrence of pharyngeal stenosis, defined by the need to perform pharyngoplasty.

SECONDARY OUTCOMES:
Delay in the occurrence of refractory stenosis or pharyngeal stenosis | at 1 month
  Time between inclusion and occurrence of refractory stenosis or pharyngeal stenosis
Delay in the occurrence of refractory stenosis or pharyngeal stenosis | at 3 months
  Time between inclusion and occurrence of refractory stenosis or pharyngeal stenosis
Delay in the occurrence of refractory stenosis or pharyngeal stenosis | at 6 months
  Time between inclusion and occurrence of refractory stenosis or pharyngeal stenosis
Delay in the occurrence of refractory stenosis or pharyngeal stenosis | at 9 months
  Time between inclusion and occurrence of refractory stenosis or pharyngeal stenosis
Delay in the occurrence of refractory esophagal stenosis or pharyngeal stenosis | at 12 months
  Time between inclusion and occurrence of refractory stenosis or pharyngeal stenosis
Distance of the stenosis | at 1 month
  Distance between the stenosis and the dental arches (cm)
Distance of the stenosis | at 3 months
  Distance between the stenosis and the dental arches (cm)
Distance of the stenosis | at 6 months
  Distance between the stenosis and the dental arches (cm)
Distance of the stenosis | at 9 months
  Distance between the stenosis and the dental arches (cm)
Distance of the stenosis | at 12 months
  Distance between the stenosis and the dental arches (cm)
Number of stenosis | at 1 month
  Number of stenosis will be evaluated by endoscopy
Number of stenosis | at 3 months
  Number of stenosis will be evaluated by endoscopy
Number of stenosis | at 6 months
  Number of stenosis will be evaluated by endoscopy
Number of stenosis | at 9 months
  Number of stenosis will be evaluated by endoscopy
Number of stenosis | at 12 months
  Number of stenosis will be evaluated by endoscopy
Length of stenosis | at 1 month
  Length of each stenosis will be evaluated by endoscopy
Length of stenosis | at 3 months
  Length of each stenosis will be evaluated by endoscopy
Length of stenosis | at 6 months
  Length of each stenosis will be evaluated by endoscopy
Length of stenosis | at 9 months
  Length of each stenosis will be evaluated by endoscopy
Length of stenosis | at 12 months
  Length of each stenosis will be evaluated by endoscopy
Estimated diameter of stenosis | at 1 month
  Diameter of each stenosis will be evaluated by endoscopy
Estimated diameter of stenosis | at 3 months
  Diameter of each stenosis will be evaluated by endoscopy
Estimated diameter of stenosis | at 6 months
  Diameter of each stenosis will be evaluated by endoscopy
Estimated diameter of stenosis | at 9 months
  Diameter of each stenosis will be evaluated by endoscopy
Estimated diameter of stenosis | at 12 months
  Diameter of each stenosis will be evaluated by endoscopy
Endoluminal inflammation | at 1 month
  Importance of endoluminal inflammation during endoscopy performed for dilation (minimal, moderate, or severe)
Endoluminal inflammation | at 3 months
  Importance of endoluminal inflammation during endoscopy performed for dilation (minimal, moderate, or severe)
Endoluminal inflammation | at 6 months
  Importance of endoluminal inflammation during endoscopy performed for dilation (minimal, moderate, or severe)
Endoluminal inflammation | at 9 months
  Importance of endoluminal inflammation during endoscopy performed for dilation (minimal, moderate, or severe)
Endoluminal inflammation | at 12 months
  Importance of endoluminal inflammation during endoscopy performed for dilation (minimal, moderate, or severe)
Number of dilation sessions | at 1 month
  Number of dilation sessions evaluated by endoscopy
Number of dilation sessions | at 3 months
  Number of dilation sessions evaluated by endoscopy
Number of dilation sessions | at 6 months
  Number of dilation sessions evaluated by endoscopy
Number of dilation sessions | at 9 months
  Number of dilation sessions evaluated by endoscopy
Number of dilation sessions | at 12 months
  Number of dilation sessions evaluated by endoscopy
Intervals between iterative dilations | at 1 month
  Time between endoscopic dilatations if necessary iterative dilation
Intervals between iterative dilations | at 3 months
  Time between endoscopic dilatations if necessary iterative dilation
Intervals between iterative dilations | at 6 months
  Time between endoscopic dilatations if necessary iterative dilation
Intervals between iterative dilations | at 9 months
  Time between endoscopic dilatations if necessary iterative dilation
Intervals between iterative dilations | at 12 months
  Time between endoscopic dilatations if necessary iterative dilation
Digestive perforations | at 1 month
  Proportion of digestive perforations secondary to endoscopic dilation
Digestive perforations | at 3 months
  Proportion of digestive perforations secondary to endoscopic dilation
Digestive perforations | at 6 months
  Proportion of digestive perforations secondary to endoscopic dilation
Digestive perforations | at 9 months
  Proportion of digestive perforations secondary to endoscopic dilation
Digestive perforations | at 12 months
  Proportion of digestive perforations secondary to endoscopic dilation
Extent of pharyngeal stenosis | at 1 month
  Laryngeal stenosis associated with pharyngeal stenosis
Extent of pharyngeal stenosis | at 3 months
  Laryngeal stenosis associated with pharyngeal stenosis
Extent of pharyngeal stenosis | at 6 months
  Laryngeal stenosis associated with pharyngeal stenosis
Extent of pharyngeal stenosis | at 9 months
  Laryngeal stenosis associated with pharyngeal stenosis
Extent of pharyngeal stenosis | at 12 months
  Laryngeal stenosis associated with pharyngeal stenosis
Proportion of unanticipated adverse reactions | at day 0
  Unanticipated adverse reactions will be defined by the occurrence of death,cardiac arrest whatever the cause,unplanned admission to intensive care unit (ICU) or extended stay > 24 ICU
Proportion of unanticipated adverse reactions | at day 2
  Unanticipated adverse reactions will be defined by the occurrence of death,cardiac arrest whatever the cause,unplanned admission to intensive care unit (ICU) or extended stay > 24 ICU
Proportion of unanticipated adverse reactions | at day 5
  Unanticipated adverse reactions will be defined by the occurrence of death,cardiac arrest whatever the cause,unplanned admission to intensive care unit (ICU) or extended stay > 24 ICU
Proportion of unanticipated adverse reactions | at day 7
  Unanticipated adverse reactions will be defined by the occurrence of death,cardiac arrest whatever the cause,unplanned admission to intensive care unit (ICU) or extended stay > 24 ICU
Proportion of unanticipated adverse reactions | at one month
  Unanticipated adverse reactions will be defined by the occurrence of death,cardiac arrest whatever the cause,unplanned admission to intensive care unit (ICU) or extended stay > 24 ICU
Proportion of unanticipated adverse reactions | at 3 months
  Unanticipated adverse reactions will be defined by the occurrence of death,cardiac arrest whatever the cause,unplanned admission to intensive care unit (ICU) or extended stay > 24 ICU
Proportion of unanticipated adverse reactions | at 6 months
  Unanticipated adverse reactions will be defined by the occurrence of death,cardiac arrest whatever the cause,unplanned admission to intensive care unit (ICU) or extended stay > 24 ICU
Proportion of unanticipated adverse reactions | at 9 months
  Unanticipated adverse reactions will be defined by the occurrence of death,cardiac arrest whatever the cause,unplanned admission to intensive care unit (ICU) or extended stay > 24 ICU
Proportion of unanticipated adverse reactions | at 12 months
  Unanticipated adverse reactions will be defined by the occurrence of death,cardiac arrest whatever the cause,unplanned admission to intensive care unit (ICU) or extended stay > 24 ICU
Proportion of adverse reactions related to corticosteroid therapy | within 7 days
  Adverse reactions related to corticosteroid therapy will be defined by the occurrence of infections needing antibiotic therapy or spontaneous digestive perforation or digestive bleeding or cardiac arrhythmias de novo or pulmonary edema requiring treatment (increased oxygen requirements and/or Diuretic and/or Vasodilator and/or non-invasive ventilation and/or invasive ventilation) or respiratory complications (High blood pressure requiring treatment - Metabolic alkalosis- Hypokalemia<3.0mmol/l - Delirium- Decompensation of a psychiatric pathology)
C-Reactive Protein (CRP) | at day 0
  Inflammation markers
C-Reactive Protein (CRP) | at day 2
  Inflammation markers
C-Reactive Protein (CRP) | at day 5
  Inflammation markers
C-Reactive Protein (CRP) | at one month
  Inflammation markers
interleukin-1 (IL1) | at day 0
  Inflammation markers
interleukin-1 (IL1) | at day 2
  Inflammation markers
interleukin-1 (IL1) | at day 5
  Inflammation markers
interleukin-1 (IL1) | at one month
  Inflammation markers
interleukin-6 (IL-6) | at day 0
  Inflammation markers
interleukin-6 (IL-6) | at day 2
  Inflammation markers
interleukin-6 (IL-6) | at day 5
  Inflammation markers
interleukin-6 (IL-6) | at one month
  Inflammation markers
Tumour Necrosis Factor alpha (TNF alpha) | at day 0
  Inflammation markers
Tumour Necrosis Factor alpha (TNF alpha) | at day 2
  Inflammation markers
Tumour Necrosis Factor alpha (TNF alpha) | at day 5
  Inflammation markers
Tumour Necrosis Factor alpha (TNF alpha) | at one month
  Inflammation markers
Tissue Growth Factor Beta (TGF beta) | at day 0
  Fibrosis markers
Tissue Growth Factor Beta (TGF beta) | at day 2
  Fibrosis markers
Tissue Growth Factor Beta (TGF beta) | at day 5
  Fibrosis markers
Tissue Growth Factor Beta (TGF beta) | at one month
  Fibrosis markers
Galectin 3 | at day 0
  Fibrosis markers
Galectin 3 | at day 2
  Fibrosis markers
Galectin 3 | at day 5
  Fibrosis markers
Galectin 3 | at one month
  Fibrosis markers

IPD SHARING:
Plan to Share IPD: Undecided